CLINICAL TRIAL: NCT00414076
Title: A Randomized Phase II Study of Letrozole Versus Observation in Patients With Newly Diagnosed Uterine Leiomyosarcoma
Brief Title: Letrozole Versus Observation in Patients With Newly Diagnosed Uterine Leiomyosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0453; NCI-2010-00554 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Leiomyosarcoma; Uterine Neoplasm
Keywords: Uterine Leiomyosarcoma; Uterine Neoplasm; Uterine Sarcomas; Uterine Cancer; Uterus; LMS; ER Positivity; Femara; Letrozole
MeSH Terms: conditions — Leiomyosarcoma; Uterine Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Active Comparator): Letrozole 2.5 mg Tablet By Mouth Daily for 12 Weeks.
  Interventions: Drug: Letrozole
- Standard of Care (No Intervention): Patients receive no treatment. Follow up every 3 months.

INTERVENTIONS:
Drug: Letrozole — 2.5 mg Tablet By Mouth Daily for 12 Weeks.
  Other Names: Femara
  Arms: Letrozole

SUMMARY:
The goal of this clinical research study is learn if taking Femara (letrozole) after a hysterectomy (surgical removal of the uterus) for uterine leiomyosarcoma will delay or prevent the cancer from coming back.

DETAILED DESCRIPTION:
Letrozole is an aromatase inhibitor. Aromatase is the enzyme that produces estrogen in post-menopausal women. By interfering with the production of estrogen triggered by aromatase, letrozole reduces the total amount of estrogen in the body. As a result, less estrogen can reach cancer cells, thus preventing their growth.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. These exams, tests, or procedures are part of regular cancer care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

Your complete medical history will be recorded, and you will have a physical exam (including a pelvic exam). Your vital signs and blood pressure will be measured. Blood (about 2-3 teaspoons) will be drawn for routine tests. You will also have a blood test (1 teaspoon) to check your cholesterol. You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart). You will also have a chest x-ray, and either a computed tomography (CT) scan or a magnetic resonance imaging (MRI) to check the status of the disease. Your doctors will test previously collected tumor tissue to learn if the estrogen receptor is positive or negative.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. Group 1 will receive letrozole by mouth once a day. Group 2 will receive no treatment. Both groups will be followed closely every 3 months. You will have an equal chance of being placed in either group.

If you are in Group 1, you will take letrozole by mouth every day for 12 weeks. Every 12 weeks is considered a study "cycle." You will only be given the amount of drug needed for 1 cycle of therapy at a time. You will keep a diary during the study that will list when and how much drug you took. This diary will be reviewed after each cycle of therapy by the research nurse or doctor and filed in your chart.

Every 12 weeks, all participants will have blood (about 3-4 teaspoons) drawn for routine tests. CT scan of the chest, abdomen (stomach area), and pelvis will be done every 24 weeks. In addition, all participants will have a physical exam (including a pelvic exam), and your vital signs and blood pressure will be measured.

You may remain on study for as long as you are benefitting. You will be taken off study if intolerable side effects occur.

Once you are off study, blood (about 2-3 teaspoons) will be drawn for routine tests and to measure your cholesterol level. You will have a physical exam (including a pelvic exam), and an MRI or CT scan.

This is an investigational study. Letrozole is approved by the FDA for treatment of some breast cancer patients after surgery. Its use in patients with leiomyosarcoma is experimental. Up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an approved informed consent.
2. Histologically confirmed uterine leiomyosarcoma with disease limited to the uterus (determined by surgical staging or radiologic imaging).
3. Tumors must express ER positivity by immunohistochemistry (ER expression >10% by immunohistochemistry).
4. Patients must have a hysterectomy and bilateral oophorectomy prior to initiation of therapy.
5. All patients must have no measurable disease. Measurable disease is defined as lesions that can be measured by physical examination or by means of imaging techniques. Imaging must be done within 6 weeks of study entry.
6. Patients must have a Zubrod performance status of 0, 1, or 2.
7. Patients must have a pretreatment granulocyte count (i.e., segmented neutrophils + bands) of greater than 1,000/Fl, a hemoglobin level of greater than or equal to 9.0 gm/dL and a platelet count of greater than 75,000/dL.
8. Patients must have an adequate renal function as documented by serum creatinine less than or equal to 2.0 mg/dL.
9. Patients must have adequate hepatic function as documented by a serum bilirubin less than or equal to 2.5 mg/dL.
10. Aspartate transaminase (SGOT) must be less than 3x institutional upper limit of normal.
11. Patients must have recovered from the effects of prior surgery.
12. No more than 12 weeks must have elapsed from hysterectomy.
13. Patients must be 18 years or older.

Exclusion Criteria:

1. Patients who do not have pure uterine sarcomas (i.e., no mixed malignant Mullerian tumors).
2. Patients with any other severe concurrent disease, which would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.
3. Patients with a history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years.
4. Patients who were taking or have a history of taking letrozole or another aromatase inhibitor.
5. Patients with active or uncontrolled systemic infection.
6. Patients with history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with an ejection fraction under 40%.
7. Patients who are pregnant or breast-feeding.
8. Presence of clinically apparent untreated central nervous system metastases.
9. Presence of carcinomatous meningitis.
10. Patients currently receiving chemotherapy or radiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-12-19 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Coleman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized (adaptive), open-label phase II of Letrozole (experimental) vs. observation (control) in patients with clinical stage I or stage II leiomyosarcoma
Pre-assignment Details: physical exam, vital signs, ECG, laboratory tests, chest x-ray, CT or MRI
Groups:
- Letrozole: Letrozole only
- Standard of Care: Standard of Care-Patients receive no treatment.
Period: Overall Study
Arm/Group | Letrozole | Standard of Care
Started | 4 | 5
Completed | 1 | 0
Not Completed | 3 | 5
Not completed — Progression | 1 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Standard of Care | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 48 [43 to 54] | 51 [38 to 60] | 49 [38 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Number of participants progressed or death from study entry.
Time Frame: Every 12 weeks
Population: 1 out of 4 participants in the Letrozole arm progressed on study. 2 participants progressed in standard of care
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Standard of Care
Number analyzed (Participants) | 4 | 5
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: From study entry to time of progression or death
Description: 5 Participants was under observation and received no treatments
Arm/Group | Letrozole | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=4) | Standard of Care (N=5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bilirubin (Metabolism and nutrition disorders) | 1 | 0
Cholesterol (Metabolism and nutrition disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Fatigue (Musculoskeletal and connective tissue disorders) | 3 | 0
Fever w/o neutropenia (General disorders) | 1 | 0
Hot Flashes (Endocrine disorders) | 4 | 0
Insomnia (General disorders) | 1 | 0
Memory Impairment (Psychiatric disorders) | 1 | 0
Mood Alteration (depression) (Psychiatric disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neuropathy: sensory (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (joint) (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (muscle) (Musculoskeletal and connective tissue disorders) | 2 | 0
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-04-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT00414076/Prot_SAP_000.pdf